CLINICAL TRIAL: NCT05681377
Title: The Impact of Administration of Flumazenil on the Emergence Delirium in Patients Anesthetized With Remimazolam: a Prospective Randomized Single-blind Study
Brief Title: Impact of Flumazenil on the Emergence Delirium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Byung Gun Lim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022GR0520
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia, General
Keywords: Remimazolam, Flumazenil, Emergence delirium, Delirium
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flumazenil group (Experimental): After discontinuation of remimazolam administration, flumazenil is administered to help the patient recover consciousness.
  Interventions: Drug: Flumazenil
- Control group (No Intervention): After discontinuation of remimazolam administration, wait until the patient's consciousness is restored naturally without flumazenil administration.

INTERVENTIONS:
Drug: Flumazenil — After cessation of remimazolam infusion, flumazenil 0.2 mg is administered intravenously over 15 seconds. If consciousness is not adequately restored within 3-5 minutes, a second dose of 0.1 mg intravenously over 15 seconds is administered. If necessary, 0.1 mg may be administered repeatedly at 3-5 minute intervals, and the maximum dose of 1 mg should not be exceeded.
  Arms: Flumazenil group

SUMMARY:
Flumazenil rapidly antagonizes benzodiazepines (BZDs); it may induce agitation, seizure, or delirium, especially when applied to patients who have taken BZDs for a long time. On the contrary, it may help patients regain consciousness in a stable and calm state by appropriately reversing the central nervous system depressant effects of BZDs. In this study, we aim to investigate the impact of flumazenil on the emergence delirium in patients anesthetized with remimazolam, the short-acting BZD drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 years or older undergoing surgery under general anesthesia

Exclusion Criteria:

* Peripheral nerve block or Neuraxial block
* Uncontrolled hypertension (HTN) (systolic blood pressure (SBP) ≥180 mmHg)
* Uncontrolled diabetes mellitus (DM) (HbA1c ≥9.0%)
* Hepatic dysfunction (Total bilirubin ≥3.0 mg/mL or Liver enzyme ≥Upper normal limit x 2.5)
* Renal dysfunction (Estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2 or Dialysis)
* Moderate or severe chronic obstructive pulmonary disease or Respiratory failure
* Emergency
* Hepatectomy or Liver transplantation
* Intraoperative cardiopulmonary bypass (CPB) or extracorporeal membrane oxygenation (ECMO) use
* Head trauma, Increased intracranial pressure, Craniotomy
* Chronic use of benzodiazepines (BZDs)
* Anxiety, Alcohol/Drug dependence, Addiction to tricyclic antidepressants (TCAs)
* Allergic reaction to BZDs, flumazenil, or other drugs used in general anesthesia
* Severe allergy or Anaphylaxis history
* Lactose-related genetic disorders
* Myasthenia gravis or Myasthenia gravis syndrome
* Myocardial infarction or Cerebrovascular events within 6 months
* Symptomatic coronary artery disease
* Organic brain disease
* Cognitive impairment (Inability to understand informed consent)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence delirium | From emergence to postanesthesia care unit (PACU) discharge (Immediately after extubation, 15 min after PACU admission, PACU discharge) [within 2 hrs after surgery]
  Richmond Agitation & Sedation Scale (RASS) ≥1 is considered emergence delirium.

SECONDARY OUTCOMES:
Incidence of postoperative delirium (POD) | From PACU to postoperative day 5(until the discharge date if discharged before 5 days after surgery) [2 times a day in the morning/afternoon]
  3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM) is used for the evaluation of POD.
Severity of POD | From PACU to postoperative day 5
  CAM-severity (CAM-S) is utilized to determine the severity of POD if it occurs.
Duration of POD | From PACU to postoperative day 5
  3D-CAM is utilized to check the duration of POD.
Level of consciousness | From emergence to PACU discharge (Immediately after extubation, 15 min after PACU admission, PACU discharge) [within 2 hrs after surgery
  Richmond Agitation & Sedation Scale (RASS) is used to evaluate the patients level of consciousness.
Incidence of resedation | From emergence to PACU discharge (Immediately after extubation, 15 min after PACU admission, PACU discharge) [within 2 hrs after surgery
  Richmond Agitation & Sedation Scale (RASS) ≤-2 is diagnosed as resedation.
Time to eye-opening | After remimazolam cessation to eye-opening [within 30 min after remimazolam cessation]
  Time taken for patients to open their eyes when their name is gently called after discontinuation of remimazolam.
Time to extubation | After remimazolam cessation to extubation [within 30 min after remimazolam cessation]
  Time taken for patients to maintain spontaneous breathing and be extubated after remimazolam discontinuation.
Preoperative anxiety | 1 day before surgery
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) is used to evaluate the patient's anxiety before surgery
Postoperative nausea/vomiting (PONV) | From immediately after extubation to PACU discharge [within 2 hours after surgery]
  Confirm PONV through patient's symptoms and signs.
Postoperative pain | From PACU admission to postoperative day 5
  Numeric rating scale (NRS) or Visual analogue scale (VAS) is used to determine the patient's pain severity (*NRS and VAS are measured on a 0-10 scale, and the higher the score, the more severe the patient's pain)
Postoperative hospital length of stay | From the day of surgery to the day of hospital discharge [within 1 month]
  Calculate the days from the date of surgery to the date of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Byung Gun Lim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
We have no plans yet to share individual participant data (IPD) with other researchers.